CLINICAL TRIAL: NCT00758576
Title: ReSTOR Natural +3.0D (Diopter) Study In Japan
Brief Title: ReSTOR Natural +3.0D Study In Japan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Kaiko Itoh, Alcon
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-07-44
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-12

CONDITIONS: Cataract
Keywords: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SN6AD1 (Experimental): AcrySof ReSTOR Model SN6AD1 Intraocular Lens
  Interventions: Device: ACRYSOF Multifocal Single-piece Intraocular Lens (IOL) Model SN6AD1

INTERVENTIONS:
Device: ACRYSOF Multifocal Single-piece Intraocular Lens (IOL) Model SN6AD1 — Implantation with the AcrySof ReSTOR Intraocular Lens (IOL) Model SN6AD1 following cataract removal.

SUMMARY:
The objective of this study is to evaluate safety and effectiveness of ACRYSOF Multifocal Single-piece Intraocular Lens (IOL) Model SN6AD1 when implanted to replace the natural lens following cataract removal.

ELIGIBILITY:
Inclusion Criteria:

* Planned bilateral cataract removal by phacoemulsification
* Potential postoperative best corrected visual acuity of 0.5 or over
* 1.5 Diopter (D) or less of astigmatism preoperatively, measured by keratometry

Exclusion Criteria:

* Poorly controlled glaucoma
* Progressive diabetic retinopathy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hayashi Eye Hospital, Fukuoka, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only adult subjects of either gender in need of cataract extraction in both eyes were considered for enrollment. 64 subjects were implanted bilaterally with the ACRYSOF® ReSTOR® Aspheric +3.0 D (Diopter) Add Power Intraocular Lens (IOL) Model SN6AD1
Pre-assignment Details: Subjects were examined to ensure inclusion/exclusion criteria. Only subjects who signed an informed consent and qualified to be in the study were enrolled. Subject numbers were assigned after obtaining consent meeting inclusion/exclusion criteria. Subjects were considered enrolled once implanted in the first operative eye.
Groups:
- SN6AD1: ACRYSOF® ReSTOR® Aspheric +3.0 D (Diopter) Add Power Intraocular Lens (IOL) Model SN6AD1
Period: Overall Study
Arm/Group | SN6AD1
Started | 64
Completed | 63
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | SN6AD1
Number analyzed (Participants) | 64
Age, Customized [Number; unit: Participants]
  <60 years of age | 6
  60 - 69 years of age | 23
  70 - 79 years of age | 33
  >80 years of age | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Intermediate Visual Acuity
Description: Binocular Uncorrected Intermediate Visual Acuity, measured at 1 meter and 50 centimeters measured in decimal visual acuity. Decimal visual acuity is the normal method to measure visual acuity in Japan. A higher decimal visual acuity value indicates better visual acuity. 0.5 in decimal visual acuity means 20/40 in Snellen fraction.
Time Frame: 1 year after surgery
Population: One patient dropped out after the visit 6 months following surgery but before the 1 year visit.
Measure: Mean (Full Range); unit: Decimal Visual Acuity
Arm/Group | SN6AD1
Number analyzed (Participants) | 63
Decimal Visual Acuity
  1 meter | 0.771 [0.3 to 1.2]
  50 centimeters | 0.861 [0.5 to 1.2]

2. Primary Outcome: Uncorrected Distance Visual Acuity
Description: Binocular Uncorrected Dinstance Visual Acuity measured in decimal visual acuity. Decimal visual acuity is the normal method to measure visual acuity in Japan. A higher decimal visual acuity value indicates better visual acuity. 0.5 in decimal visual acuity means 20/40 in Snellen fraction.
Time Frame: 1 year after surgery
Population: One patient dropped out after the visit 6 months following surgery but before the 1 year visit.
Measure: Mean (Full Range); unit: Decimal Visual Acuity
Arm/Group | SN6AD1
Number analyzed (Participants) | 63
Decimal Visual Acuity | 1.122 [0.4 to 2.0]

3. Primary Outcome: Uncorrected Near Visual Acuity
Description: Binocular Near Visual Acuity measured in decimal visual acuity. Decimal visual acuity is the normal method to measure visual acuity in Japan. A higher decimal visual acuity value indicates better visual acuity. 0.5 in decimal visual acuity means 20/40 in Snellen fraction.
Time Frame: 1 year after surgery
Population: One patient dropped out after the visit 6 months following surgery but before the 1 year visit.
Measure: Mean (Full Range); unit: Decimal Visual Acuity
Arm/Group | SN6AD1
Number analyzed (Participants) | 63
Decimal Visual Acuity | 1.082 [0.6 to 1.9]

ADVERSE EVENTS:
Time Frame: From time of surgery to 1 year following surgery.
Arm/Group | SN6AD1
Serious Adverse Events (participants affected / at risk) | 1/64
Other Adverse Events (participants affected / at risk) | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SN6AD1 (N=64)
Stroke (Nervous system disorders) | 1 (1) — No causality with the test article

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less